CLINICAL TRIAL: NCT05672485
Title: 99mTc-P137 SPECT/CT Molecular Probe in Precise Diagnosis of Prostate Cancer
Brief Title: 99mTc-P137 SPECT/CT in Prostate Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: XJTU1AF2022LSK-356
Record Dates: First submitted 2023-01-03; First posted 2023-01-05 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2022-12

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients diagnosed with prostate cancer (Experimental)
  Interventions: Diagnostic Test: SPECT/CT imaging with 99mTc-P137 nuclide probe

INTERVENTIONS:
Diagnostic Test: SPECT/CT imaging with 99mTc-P137 nuclide probe — inject the tracer 99mTc-P137 to subjects and perform SPECT/CT scans

SUMMARY:
Purpose: This study will take prostate specific membrane antigen (PSMA) as the targeting of radionuclide labeled molecular probe to explore the diagnostic efficacy of 99mTc-P137 radioactive probe in prostate cancer. Combining with SPECT/CT to optimize the imaging, image analysis and clinical diagnosis process of 99mTc-P137 probe, the aim of the study is to provide new methods and new means for the early detection, early diagnosis, accurate tumor staging, treatment decision and prognosis judgment of malignant tumor, and will provide scientific and clinical basis for the precise diagnosis and treatment of prostate cancer.

Research objectives: To investigate the clinical translational application value of 99mTc-P137 molecular probe in accurate detection of prostate cancer lesions.

Research design: A prospective study design will be used in this study. Patients meeting the inclusion criteria of this study will be analyzed with 99mTc-P137 SPECT/CT imaging. To evaluate the diagnostic and prognostic value of 99mTc-P137 nuclear medicine imaging in accurate detection of prostate cancer lesions, clinical surgical specimens and pathological diagnosis will be used as the gold standard.

Study the population Indications: For patients with suspected prostate cancer who plan to undergo surgical resection or puncture biopsy after various examinations, the final pathological results can be obtained.

ELIGIBILITY:
Inclusion Criteria:

* patients age 18 or above;
* highly suspicious for prostate cancer patients: 1) Serum PSA is significantly changed compared with before (PSA<4.0ng/mL with annual change >0.35ng/mL; or PSA > 4.0ng/mL with annual change > 0.75ng/mL); 2) First or second degree relatives have a history of prostate cancer; 3) Nuclear magnetic PI-RADS score ≥3 points;
* the prostate biopsy or surgical pathology is diagnosed with prostate cancer;
* available to provide clinical laboratory results (blood routine, biochemical and serum PSA) within one month before this study; At least two imaging examinations including CT, MRI, nuclear medicine (PET/CT or SPECT/CT), ultrasound and other imaging techniques;
* Can complete the inspection autonomously;
* voluntary and signed informed consent.

Exclusion Criteria:

* there are other malignant tumor history;
* severe damage of liver and kidney function;
* may not be able to obtain pathology or long-term follow-up results;
* don't have access to relevant reference image data and clinical data;
* difficult to cooperate.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-01-05 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
99mTc-P137 SPECT/CT imaging | 2 hours after injection
  Qualitative and semi-quantitative analysis (T/N ratio of tumor lesion and adjacent normal tissue, changes in uptake of lesion of interest before and after treatment, and early and late imaging)

SECONDARY OUTCOMES:
Other imaging findings | 7 days with the injection
  CT, PET/CT, SPECT/CT and MRI will be used to evaluate the lesion scope, size and metastasis of the tumor

CONTACTS AND LOCATIONS:
Overall Officials: Rui Gao, Study Chair — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol